CLINICAL TRIAL: NCT01195675
Title: Assessment of the Effect of 25 mg and 200 mg of BI 10773 as Single Dose on the QT Interval in Healthy Female and Male Subjects. A Randomised, Placebo Controlled, Double-blind, Five-period Crossover Phase-I-study With Moxifloxacin as Positive Control
Brief Title: Assessment of the Effect of Empagliflozin (BI 10773) as Single Dose on the QT Interval in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.16; 2010-018609-13 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Moxifloxacin

ARMS (3):
- BI 10773 (Experimental): single oral (high and low) dose per subject
  Interventions: Drug: BI 10773 (low); Drug: BI 10773 (high)
- Placebo (Placebo Comparator): 2 single oral doses per subject
  Interventions: Drug: BI 10773 Placebo
- Moxifloxacin (Active Comparator): single oral dose per subject
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: BI 10773 (low) — single oral dose
  Arms: BI 10773
Drug: Moxifloxacin — single oral dose
  Arms: Moxifloxacin
Drug: BI 10773 Placebo — 2 times single dose
  Arms: Placebo
Drug: BI 10773 (high) — single oral dose
  Arms: BI 10773

SUMMARY:
The objective of this study is to demonstrate that BI 10773 does not prolong the QT(c) interval more than placebo

ELIGIBILITY:
Inclusion criteria:

healthy female and male subjects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.16.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Ring A, Brand T, Macha S, Breithaupt-Groegler K, Simons G, Walter B, Woerle HJ, Broedl UC. The sodium glucose cotransporter 2 inhibitor empagliflozin does not prolong QT interval in a thorough QT (TQT) study. Cardiovasc Diabetol. 2013 Apr 24;12:70. doi: 10.1186/1475-2840-12-70. PMID 23617452

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Overall: Total number of patients randomised and treated in the study. This was a randomised, placebo controlled, 5-period crossover trial, participants were randomised to one of ten possible treatment sequences. The treatments administered were
  * 25mg empa administered orally on day 1 of the treatment period
  * 200mg empa administered orally on day 1 of the treatment period
  * 400mg moxifloxacin administered orally on day 1 of the treatment period
  * Placebo 1 administered orally on day 1 of the treatment period
  * Placebo 2 administered orally on day 1 of the treatment period
  The trial was double-blind for the placebo and Empagliflozin (Empa) treatments, but open-label for the moxifloxacin treatment. A washout period of at least 1 week was respected between drug administrations.
Period: Overall Study
Arm/Group | Study Overall
Started | 30
Received Empa 25mg | 28
Received Empa 200mg | 30
Received Moxifloxacin | 29
Received Placebo 1 | 29
Received Placebo 2 | 28
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: Total number of patients randomised and treated in the study.
Arm/Group | Study Overall
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Empa 25mg: Mean QTcN Change From Baseline Between 1 and 4 Hours After Dosing
Description: Mean QTcN (heart rate-corrected QT interval, using a study population-based approach) from the ECGs obtained between 1h to 4h following drug administration minus the mean QTcN from the baseline electrocardiogram (ECGs) obtained pre-dose at each visit, for empa 25mg.
  Note, the treatment means presented are actually adjusted means.
Time Frame: 60 minutes (min), 50min and 40 min before the first dose and 1 hour (h), 1.5h, 2h, 2.5h, 3h and 4h after the first dose
Population: Full analysis set (FAS): all treated subjects who had at least one baseline assessment and at least one post-baseline assessment for at least one ECG endpoint.
Measure: Mean (Standard Error); unit: ms
Units Other Than Participants: Observations
Groups:
- Placebo: Single oral dose of placebo (8 tablets).
- Empa 25 mg: Single oral dose of Empagliflozin (Empa) 25mg (1 tablet with strength 25mg) plus 7 tablets of placebo.
Arm/Group | Placebo | Empa 25 mg
Number analyzed (Participants) | 29 | 28
Number analyzed (Observations) | 57 | 28
ms | 3.68 (1.00) | 4.27 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Empa 25 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo; ANCOVA; Based on ANCOVA with terms for sequence, subjects within sequence, period, treatment and baseline; Mean Difference (Final Values) = 0.59, 90% CI 2-sided [-0.69 to 1.87], Standard Error of Mean 0.76 — Mean difference = Empa minus placebo

2. Secondary Outcome: Empa 25 mg: Mean QTcN Change From Baseline Between 30 Minutes and 24 Hours After Dosing
Description: Mean changes from baseline in QTcN from all ECGs taken between 30 minutes and 24 hours after dosings, for empa 25 mg.
  Note, presented means are actually adjusted means.
Time Frame: 60 minutes (min), 50min and 40 min before the first dose and 30min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after the first dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ms
Units Other Than Participants: Observations
Arm/Group | Placebo | Empa 25 mg
Number analyzed (Participants) | 29 | 28
Number analyzed (Observations) | 57 | 28
ms | 0.71 (0.99) | 1.37 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Empa 25 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo. Non-confirmatory testing; ANCOVA; Based on ANCOVA with terms for sequence, subjects within sequence, period, treatment and baseline; Mean Difference (Final Values) = 0.66, 90% CI 2-sided [-0.38 to 1.71], Standard Error of Mean 0.62 — Mean difference = Empa minus placebo

3. Secondary Outcome: Empa 200 mg: Mean QTcN Change From Baseline Between 30 Minutes and 24 Hours After Dosing
Description: Mean changes from baseline in QTcN from all ECGs taken between 30 minutes and 24 hours after dosings, for empa 200 mg.
  Note, presented means are actually adjusted means.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Units Other Than Participants: Observations
Groups:
- Empa 200 mg: Single oral dose of Empagliflozin (Empa) 200 mg (consisting of 8 tablets with strength 25 mg)
Arm/Group | Placebo | Empa 200 mg
Number analyzed (Participants) | 29 | 30
Number analyzed (Observations) | 57 | 30
ms | 0.68 (0.80) | 0.53 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Empa 200 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo. Non-confirmatory testing; ANCOVA; Based on ANCOVA with terms for sequence, subjects within sequence, period, treatment and baseline; Mean Difference (Final Values) = -0.15, 90% CI 2-sided [-1.23 to 0.93], Standard Error of Mean 0.65 — Mean difference = Empa minus placebo

4. Secondary Outcome: Mean QTcN Change From Baseline Between 2 and 4 Hours After Dosing
Description: Mean changes from baseline in QTcN from all ECGs taken between 2 hours and 4 hours after dosings
  Note, the means presented are actually adjusted means.
Time Frame: 60 minutes (min), 50min and 40 min before the first dose and 2 hour (h), 2.5h, 3h and 4h after the first dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ms
Units Other Than Participants: Observations
Groups:
- Moxifloxacin: Single oral dose of moxifloxacin 400 mg (1 tablet)
Arm/Group | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 29
Number analyzed (Observations) | 57 | 29
ms | 3.53 (1.10) | 15.96 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Moxifloxacin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on ANCOVA with terms for treatment, period, treatment sequence, baseline and subject within sequence; Mean Difference (Final Values) = 12.42, 90% CI 2-sided [10.73 to 14.11], Standard Error of Mean 1.01 — Non-confirmatory testing. Mean difference = Moxifloxacin minus placebo

5. Secondary Outcome: Empa 25mg: Change From Mean Baseline in QTcN at Each Time Point Between 30 Minutes and 24 Hours After Dosings
Description: Change from mean baseline in QTcN at each time point between 30 minutes and 24 hours after dosings for empa 25mg. The clinically relevant information (and endpoint resulting from ICH E14) is shown by the maximum upper confidence limit value over time.
  For this outcome results are presented for the 24 hour timepoint as this was when the maximum value was seen.
  Note, the presented means are actually adjusted means.
Time Frame: 60 minutes (min), 50min and 40 min before the first dose and 0.5 hour (h), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after the first dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ms
Units Other Than Participants: Observations
Arm/Group | Placebo | Empa 25 mg
Number analyzed (Participants) | 29 | 28
Number analyzed (Observations) | 57 | 28
ms | -4.46 (0.96) | -2.30 (1.30)
Statistical Analysis 1: Comparison: Placebo vs Empa 25 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo. Non-confirmatory testing; Repeated measures analysis; Based on repeated measured analysis with terms for subject, baseline, period, treatment, time, baseline by time, period by time and treatment by time; Mean Difference (Final Values) = 2.16, 90% CI 2-sided [-0.34 to 4.67], Standard Error of Mean 1.50 — Mean difference = Empa minus placebo

6. Secondary Outcome: Empa 200mg: Change From Mean Baseline in QTcN at Each Time Point Between 30 Minutes and 24 Hours After Dosings
Description: Change from mean baseline in QTcN at each time point between 30 minutes and 24 hours after dosings for empa 200mg. The clinically relevant information (and endpoint resulting from ICH E14) is shown by the maximum upper confidence limit value over time.
  For this outcome results are presented for the 2.5 hour timepoint as this was when the maximum value was seen.
  Note, the presented means are actually adjusted means.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ms
Units Other Than Participants: Observations
Arm/Group | Placebo | Empa 200 mg
Number analyzed (Participants) | 29 | 30
Number analyzed (Observations) | 57 | 30
ms | 3.05 (0.96) | 4.64 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Empa 200 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo. Non-confirmatory testing; Repeated measures analysis; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 1.59, 90% CI 2-sided [-0.35 to 3.53], Standard Error of Mean 1.16 — Mean difference = Empa minus placebo

7. Primary Outcome: Empa 200mg: Mean QTcN Change From Baseline Between 1 and 4 Hours After Dosing
Description: Mean QTcN (heart rate-corrected QT interval, using a study population-based approach) from the ECGs obtained between 1h to 4h following drug administration minus the mean QTcN from the baseline ECGs obtained pre-dose at each visit, for empa 200mg.
  Note, the treatment means presented are actually adjusted means.
Time Frame: 60 minutes (min), 50min and 40 min before the first dose and 1 hour (h), 1.5h, 2h, 2.5h, 3h and 4h after the first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Units Other Than Participants: Observations
Arm/Group | Placebo | Empa 200 mg
Number analyzed (Participants) | 29 | 30
Number analyzed (Observations) | 57 | 30
ms | 3.67 (0.86) | 3.44 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Empa 200 mg; Non-inferiority margin: 10ms; Test type: Non-Inferiority or Equivalence — Empa vs placebo; ANCOVA; Based on ANCOVA with terms for sequence, subjects within sequence, period, treatment and baseline; Mean Difference (Final Values) = -0.22, 90% CI 2-sided [-1.39 to 0.94], Standard Error of Mean 0.69 — Mean difference = Empa minus placebo

8. Other Pre Specified Outcome: Time-matched Change From Placebo in QTcN Between 30 Minutes and 24 Hours After Dosing.
Description: The time-matched change from placebo is defined per time point as the difference of the ECG measurement following administration of empa or moxifloxacin minus the average of the measurements obtained following the two administrations of placebo. The clinically relevant information (and endpoint resulting from ICH E14) is shown by the maximum mean value of all measurements.
  Results are presented for the greatest change, for empa 25mg the greatest change was seen at the 24 hour time point, for empa 200 mg and moxifloxacin the greatest change was seen at the 2.5 hour time point.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Empa 25 mg: Single oral dose of Empagliflozin (Empa) 25mg (1 tablet) plus 7 tablets of placebo.
Arm/Group | Empa 25 mg | Empa 200 mg | Moxifloxacin
Number analyzed (Participants) | 28 | 29 | 29
ms | 4.05 (5.62) | 3.45 (10.18) | 13.99 (8.19)

9. Other Pre Specified Outcome: Placebo Corrected Change From Mean Baseline at Any Time Point Between 30 Minutes and 24 Hours After Dosings.
Description: The placebo corrected change from mean baseline is defined per time point as the difference of the change from baseline for empa or moxifloxacin minus the average change from baseline obtained for the two administrations of placebo. The clinically relevant information (and endpoint resulting from ICH E14) is shown by the maximum mean value of all measurements.
  Results are presented for the greatest change, for empa 25mg the greatest change was seen at the 24 hour time point, for empa 200 mg and moxifloxacin the greatest change was seen at the 2.5 hour time point.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Empa 200 mg: Single oral dose of Empagliflozin (Empa) 200 mg (8 tablets of 25 mg)
Arm/Group | Empa 25 mg | Empa 200 mg | Moxifloxacin
Number analyzed (Participants) | 28 | 29 | 29
ms | 1.70 (7.64) | 1.67 (8.48) | 13.43 (8.38)

10. Other Pre Specified Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Assessment of Tolerability by the Investigator
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, blood chemistry, haematology, urinanalysis and assessment of tolerability by the investigator. New abnormal findings or worsening of baseline conditions were reported as adverse events (AEs). Time frame for AE reporting includes the period of first drug administration until end of study. A more detailed definition of the used time frame and MedDRA Version can be found in the AE section.
Time Frame: Drug administration until beginning of next sequence/end of trial, up to 48 days
Population: Treated set (TS): All subjects who were dispensed trial medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 25 mg | Empa 200 mg | Moxifloxacin
Number analyzed (Participants) | 29 | 28 | 30 | 29
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Drug administration until beginning of next sequence/end of trial, up to 48 days
Arm/Group | Placebo | Empa 25 mg | Empa 200 mg | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/30 | 1/29
Other Adverse Events (participants affected / at risk) | 6/29 | 3/28 | 2/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Empa 25 mg (N=28) | Empa 200 mg (N=30) | Moxifloxacin (N=29)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Empa 25 mg (N=28) | Empa 200 mg (N=30) | Moxifloxacin (N=29)
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.